CLINICAL TRIAL: NCT02773914
Title: Comprehensive Geriatric Assessment for Frail Older People in Swedish Acute Care Settings: A Randomized Controlled Study
Brief Title: Comprehensive Geriatric Assessment for Frail Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CGA for frail older people
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Dependency
Keywords: Activity of Daily Living (ADL); Comprehensive Geriatric Assessment; Elderly; Frailty; Randomized controlled study
MeSH Terms: conditions — Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CGA intervention (Experimental): The CGA intervention will include multidisciplinary teams consisting of physician, nurse (RN), physiotherapist (PT), occupational therapist (OT) and social worker (SW). The team will work according to CGA, and have the primary and continuing responsibility for planning of hospital care and discharge. CGA will include assessment of socio-demographic background, social network, health and medical history, medications, functional status, cognitive status, nutritional status, somatic status and psychosocial status including depression, as well as treatment and planning for discharge and follow-up.
  Interventions: Other: Comprehensive Geriatric Assessment
- Control group (No Intervention): The control group receives usual hospital care, that is care given at an ordinary medical hospital ward, without the specialized multi-disciplinary team approach and CGA.

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Comprehensive Geriatric Assessment intervention
  Arms: CGA intervention

SUMMARY:
The study "Comprehensive Geriatric Assessment for frail older people in Swedish acute care settings - a randomized controlled study" comprised two study arms: one intervention and one control group. The aim of the study was to evaluate the effects of the Comprehensive Geriatric Assessment (CGA) for frail older people in Swedish acute hospital settings - the CGA-Swed study. The intervention group received the CGA and a control group received medical assessment without the CGA. Follow-ups were conducted after 1, 6 and 12 months, with dependence in activities of daily living (ADL) as the primary outcome measure. The study group consisted of frail older people, 75 years and older, in need of acute medical hospital care. The study design, randomization and process evaluation carried out were intended to ensure the quality of the study. Baseline data showed that the randomisation was successful and that the sample included frail older people with high dependence in ADL, and with a high comorbidity. Thus, the CGA contributed to early recognition of frail older people's needs and ensured a care plan and follow-up. When investigating the long-term effects on frail older people's ADL 12 months after receiving the CGA, results showed that twelve participants in the intervention group (15.4%), and four participants in the control group (5.2%) had improved in their ADL 1 year after discharge. Qualitative interviews with CGA-participants also showed that the participants felt respected as a person when receiving care on a CGA acute geriatric ward.

DETAILED DESCRIPTION:
The aim of the study "Comprehensive Geriatric Assessment for frail older people in Swedish acute care settings - a randomized controlled study" was to evaluate the effects of the Comprehensive Geriatric Assessment (CGA) for frail older people in Swedish acute hospital settings.

The study addressed the following research questions:

1. Can Comprehensive Geriatric Assessment for frail older patients in Swedish acute hospital settings:

   * increase/maintain independence, functional status, health related quality of life and life satisfaction?
   * increase satisfaction with health care?
   * reduce health care consumption?
2. How feasible and acceptable are the study processes and procedures of CGA from the perspective of care givers and older persons in Swedish settings?

The intervention addressed people 75 years and older who were seeking acute hospital care at the hospital emergency department, and who were identified as being frail. The CGA intervention included a multidisciplinary team that assessed the patient's socio-demographic background, social network, health and medical history, medications, functional status, cognitive status, nutritional status, somatic status and psychosocial status including depression, as well as treatment and planning for discharge and follow-up. The intervention was person-centred, and comprised a comprehensive assessment tailored for each person.

In total, one-hundred and fifty-five people participated in the study; 78 in the intervention group and 77 in the control group. Participants in the intervention group had a higher odds ratio of reporting having received written information and felt that care met their needs during their hospital stay. At the 12-month follow up, 78 people participated (40 in the control and 38 in the intervention). Results showed that twelve participants in the intervention group (15.4%), and four participants in the control group (5.2%) had improved in their ADL 1 year after discharge. Further, people who received the CGA intervention had higher odds of receiving antidepressant treatment, suggesting that CGA improves recognition of mental health needs during an unplanned hospital admission. Qualitative interviews with participants receiving the CGA showed that the care they received on the CGA ward met their needs. The participants felt respected as a person when receiving care on a CGA acute geriatric ward. This was achieved by having a reciprocal relationship with the ward staff, enabling their participation in decisions when engaged in communication and understanding.

ELIGIBILITY:
Inclusion Criteria:

* All patients 75 years and older seeking acute hospital care at the hospital emergency department will be screened for frailty.

Exclusion Criteria:

* Those with symptoms of predefined diagnoses such as stroke, acute myocardial infarction and hip fractures, admitted through "fast tracks" directly to a designated ward without passing the emergency department.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Andersson Hammar, Assoc.prof, Principal Investigator — Göteborg University; Katarina Wilhelmson, Professor, Study Director — Göteborg University
Locations (1):
- Isabelle Andersson Hammar, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andersson Hammar I, Westgard T, Dahlin-Ivanoff S, Wilhelmson K. Frail older people with decreased cognition can perceive reduced self-determination in self-care and social relationships. BMC Geriatr. 2024 Jan 3;24(1):7. doi: 10.1186/s12877-023-04492-y. PMID 38172750
- [Result] Westgard T, Hammar IA, Wilhelmson K, Waern M. Comprehensive geriatric assessment is associated with increased antidepressant treatment in frail older people with unplanned hospital admissions-results from the randomised controlled study CGA-Swed. BMC Geriatr. 2022 Aug 5;22(1):645. doi: 10.1186/s12877-022-03324-9. PMID 35931975
- [Result] Wilhelmson K, Andersson Hammar I, Westgard T, Holmquist Henrikson L, Dahlin-Ivanoff S. Positive effects on activities of daily living one year after receiving comprehensive geriatric assessment - results from the randomised controlled study CGA-Swed. BMC Geriatr. 2022 Mar 3;22(1):180. doi: 10.1186/s12877-022-02862-6. PMID 35240988
- [Result] Wilhelmson K, Hammar IA, Ehrenberg A, Niklasson J, Eckerblad J, Ekerstad N, Westgard T, Holmgren E, Aberg ND, Ivanoff SD. Comprehensive Geriatric Assessment for Frail Older People in Swedish Acute Care Settings (CGA-Swed): A Randomised Controlled Study. Geriatrics (Basel). 2020 Jan 24;5(1):5. doi: 10.3390/geriatrics5010005. PMID 31991598
- [Result] Westgard T, Andersson Hammar I, Dahlin-Ivanoff S, Wilhelmson K. Can Comprehensive Geriatric Assessment Meet Frail Older People's Needs? Results from the Randomized Controlled Study CGA-Swed. Geriatrics (Basel). 2020 Dec 4;5(4):101. doi: 10.3390/geriatrics5040101. PMID 33291834
- [Result] Westgard T, Wilhelmson K, Dahlin-Ivanoff S, Ottenvall Hammar I. Feeling Respected as a Person: a Qualitative Analysis of Frail Older People's Experiences on an Acute Geriatric Ward Practicing a Comprehensive Geriatric Assessment. Geriatrics (Basel). 2019 Jan 25;4(1):16. doi: 10.3390/geriatrics4010016. PMID 31023984
- [Result] Westgard T, Ottenvall Hammar I, Holmgren E, Ehrenberg A, Wisten A, Ekdahl AW, Dahlin-Ivanoff S, Wilhelmson K. Comprehensive geriatric assessment pilot of a randomized control study in a Swedish acute hospital: a feasibility study. Pilot Feasibility Stud. 2018 Jan 29;4:41. doi: 10.1186/s40814-018-0228-1. eCollection 2018. PMID 29423259

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CGA Intervention | Control Group
Started | 78 | 77
Completed | 38 | 40
Not Completed | 40 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGA Intervention | Control Group | Total
Number analyzed (Participants) | 78 | 77 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 78 | 77 | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 31 | 34 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants] | 78 | 77 | 155

OUTCOME MEASURES:

1. Primary Outcome: Dependence in Activities of Daily Living
Description: Changes in number of person dependent in one or more daily activity from baseline to follow-up.
  Dependence in daily activities was measured using the ADL-staircase assessment by combining both interviews and observations. It includes dependence in nine activities: cleaning, shopping, transportation, cooking, bathing, dressing, going to the toilet, transferring and feeding. Dependence was defined as a state in which another person is involved in the activity by giving personal or directive assistance. The sum of dependence in the nine activities of daily living is calculated, range 0-9, with a clinically significant change of ≥1 unit between baseline and follow-up. At baseline, personal ADL (PADL: bathing, dressing, going to the toilet, transferring and feeding) was inquired for both actual PADL status during the hospital stay and retrospectively for PADL before onset of the acute illness leading to the hospital admission.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | CGA Intervention | Control Group
Number analyzed (Participants) | 78 | 77
Participants | 78 | 77

2. Secondary Outcome: Self-rated Health
Description: Changes in number of person with good self-rated health from baseline to follow-up.
  Self-rated health was measured by the question: "In general, would you say your health is", with the response alternatives: excellent, very good, good, fair, and poor. Clinically significant difference was defined as ≥1 step in the response alternatives between baseline and follow-up.
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2024-12

3. Secondary Outcome: Satisfaction With Quality of Care
Description: Satisfaction of care scored on a five answer statements using a likert-scale. Satisfaction with quality of care was measured by the participant's agreement with six statements with a person-centred approach: "I feel that the care given during the hospital stay meets my needs", "I feel that the care planning meeting before discharge was valuable", "I was able to take part in the discussion of my needs in the care planning meeting", "I feel that the actions planned equal my needs", "I feel that the actions delivered equal my needs" and "I am satisfied with the hospital care". The response alternatives were agree completely, agree partly, neither agree nor disagree, disagree, and disagree completely. An answer of agree completely or agree partly were considered as satisfied. These questions were only measured once (at 1 month follow-up) and were used as the difference between intervention and control groups in the proportion of participants being satisfied for each question at follow-up
Time Frame: 1 month follow-up
Reporting Status: Not Posted, anticipated posting 2024-12

4. Secondary Outcome: Life Satisfaction
Description: Life satisfaction was measured using the Fugl-Meyer-Lisat-11 Questionnaire which includes 11 items concerning satisfaction with: life as a whole, work, financial situation, leisure, friends and acquaintances, sexual life, functional capacity, family life, partner relationship, physical health and psychological health. Response alternatives included: very dissatisfied, dissatisfied, rather dissatisfied, rather satisfied, satisfied and very satisfied. In the analysis, the responses to each question were dichotomised into satisfied (very satisfied and satisfied) or not satisfied (rather satisfied, rather dissatisfied, dissatisfied and very dissatisfied) as was done in the validation of the questionnaire. The sum of items for which the respondent reported being satisfied were calculated, range 0-11, with a clinically significant change of ≥1 between baseline and follow-up.
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 3, 6 and 12 months.
Arm/Group | CGA Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/77
Other Adverse Events (participants affected / at risk) | 0/78 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT02773914/Prot_SAP_000.pdf